CLINICAL TRIAL: NCT04509622
Title: An Expanded Access Study for Venetoclax in Combination With Low-Dose Cytarabine in Treatment-Naïve Subjects With Acute Myeloid Leukemia Who Are Ineligible for Intensive Induction Therapy in Japan
Brief Title: A Study of Oral Venetoclax Tablet in Combination With Subcutaneous Low-Dose Cytarabine (LDAC) Injection to Assess Adverse Events in Adult Japanese Participants With Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M19-916
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Acute Myeloid Leukemia (AML); Cancer; Venetoclax, Venclexta
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms | interventions — venetoclax; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Venetoclax + Low-Dose Cytarabine (LDAC) (Experimental): Participants will receive venetoclax once daily (QD) on days 1 through 28 plus LDAC QD on days 1 through 10 during the 28-day treatment cycles.
  Interventions: Drug: Venetoclax; Drug: Cytarabine

INTERVENTIONS:
Drug: Venetoclax — Tablet; Oral
  Other Names: ABT-199; Venclexta
Drug: Cytarabine — Subcutaneous Injection

SUMMARY:
Acute Myeloid Leukemia (AML) is a cancer of the white blood cells which perform many functions, including fighting bacterial infections and defending the body against parasites. This study will evaluate how safe venetoclax is and assess the adverse events in adult participants with AML.

Venetoclax in combination with low-dose cytarabine (LDAC) is an approved therapy in the United States for patients with newly diagnosed acute myeloid leukemia (AML) aged > 18 years with a medical condition that prevents the use of intensive chemotherapy. This study provides access to venetoclax in combination with LDAC to participants over 18 years who are ineligible for intensive induction therapy. Around 38 adult participants with diagnosis of AML will be enrolled in approximately 15 sites across Japan.

Participants will receive oral venetoclax tablets once daily on days 1-28 in combination with subcutaneous low-dose cytarabine (LDAC) injections once daily on days 1-10 of the 28-day treatment cycles.

Participants will attend regular visits during the study at a hospital to evaluate safety by medical assessments and blood tests.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of AML, previously untreated, ineligible for intensive induction regimen due to age or co-morbidities.
* Participants who are >= 75 years of age or who are >= 18 to 74 years of age with at least one of the following co-morbidities:

  * Eastern Cooperative Oncology Group (ECOG) performance status of 2 or 3.
  * Cardiac history of congestive heart failure requiring treatment or ejection fraction <= 50% or chronic stable angina.
  * Diffusion capacity of lung for carbon monoxide (DLCO) <= 65% or forced expiratory volume during the first second (FEV1) <= 65%.
  * Adequate renal and hepatic criteria as described in the protocol.
  * Other co-morbidities that the physician judges to be incompatible with intensive chemotherapy must be reviewed and approved by the AbbVie Therapeutic Area Medical Director (TA MD) before study enrollment.

Exclusion Criteria:

* History of prior treatment for AML with the exception of hydroxyurea, allowed through the first cycle of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to approximately 9 months after the first participant receives first dose of study drug
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (16):
- Japan (16):
  - NHO Nagoya Medical Center /ID# 223671, Nagoya, Aichi-ken
  - Aichi Cancer Center Hospital /ID# 223134, Nagoya, Aichi-ken
  - University of Fukui Hospital /ID# 223133, Yoshida-gun, Fukui
  - Kyushu University Hospital /ID# 223136, Fukuoka, Fukuoka
  - Gunmaken Saiseikai Maebashi Hospital /ID# 223301, Maebashi, Gunma
  - National Hospital Organization Mito Medical Center /ID# 223392, Higashi Ibaraki-gun, Ibaraki
  - Hitachi General Hospital /ID# 223084, Hitachi-shi, Ibaraki
  - University Hospital Kyoto Prefectural University of Medicine /ID# 223135, Kyoto, Kyoto
  - Tohoku University Hospital /ID# 223169, Sendai, Miyagi
  - Okayama University Hospital /ID# 222990, Okayama, Okayama-ken
  - Osaka City University Hospital /ID# 224269, Osaka, Osaka
  - Saitama Medical University International Medical Center /ID# 223575, Hidaka-shi, Saitama
  - Juntendo University Hospital /ID# 223086, Bunkyo-ku, Tokyo
  - The Jikei University Daisan Hospital /ID# 223418, Komae-shi, Tokyo
  - NTT Medical Center Tokyo /ID# 223574, Shinagawa-ku, Tokyo
  - Yamagata University Hospital /ID# 223032, Yamagata, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=M19-916&Latitude=&Longitude=&LocationName=#additional-resources-section